CLINICAL TRIAL: NCT03902691
Title: A Phase 3, Randomized, Open-Label, Active-Controlled, Multicenter, Non-Inferiority Study to Evaluate the Efficacy and Safety of Pegol-Sihematide for Anemia in Patients With Chronic Kidney Disease on Dialysis
Brief Title: Study of the Efficacy and Safety of Pegol-Sihematide for Anemia in Patients With Chronic Kidney Disease on Dialysis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Jiangsu Hansoh Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HS-20039-302
Record Dates: First submitted 2019-03-13; First posted 2019-04-04 (Actual); Last update posted 2023-03-09 (Actual); Status verified 2022-02

CONDITIONS: Chronic Kidney Diseases
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pegol-Sihematide (Experimental): Participants received Pegolsihematide by intravenous injection once every 4 weeks.
  Interventions: Drug: Pegol-Sihematide
- ESPO (Recombinant Human Erythropoietin Injection） (Active Comparator): ESPO administration 1 to 3 times per week.
  Interventions: Drug: ESPO

INTERVENTIONS:
Drug: Pegol-Sihematide — Participants received Pegol-Sihematide by subcutaneous injection once every 4 weeks ; the dose was adjusted throughout the study to maintain a hemoglobin target range of 10.0-12.0 grams per deciliter (g/dL).
  Arms: Pegol-Sihematide
Drug: ESPO — Participants received ESPO by subcutaneous injection or subcutaneous injection weekly. The dose was adjusted throughout the study to maintain a hemoglobin target range of 10.0-12.0 g/dL.
  Arms: ESPO (Recombinant Human Erythropoietin Injection）

SUMMARY:
The purpose of this study is to evaluate the effecacy and safety of dialysis centers switching its dialysis patients from using recombinant human erythropoietin injection (CHO Cell) (ESPO) to Pegol-Sihematide injection on hemoglobin levels and other parameters.

DETAILED DESCRIPTION:
This is a phase 3, randomized, multicenter, open-label, active-controlled, non-inferiority trial to evaluate the efficacy and safety of from ESPO to monthly Pegol-Sihematide injection for the treatment of anemia in participants with chronic kidney disease（CKD）, who are on maintenance dialysis. Study included a period of 4 weeks for screening, 8 weeks for baseline, 16 weeks for dose adjustment, 8 weeks for evaluation, and 28 weeks for extensional treatment period. All patients who passed the screening were received ESPO in baseline period, then, eligible patients were centrally allocated in a 2:1 ratio to receive Pegol-Sihematide or ESPO. Doses of both drugs were adjusted to achieve and maintain hemoglobin levels between 10.0 and 12.0 g per deciliter for 52 weeks or more. The primary efficacy end point was the mean change from the baseline hemoglobin level to the mean level during the evaluation period; non-inferiority was established if the lower limit of the two-sided 95% confidence interval was -1.0 g per deciliter or higher. Cardiovascular safety was evaluated on the basis of an adjudicated composite end point.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must meet all of the following inclusion criteria to be eligible for participation in this study:

  1. Males or females ≥18 and ≤70 years of age, weight ≥ 45 kilograms (kg).
  2. Females of child-bearing potential who are sexually active had to be willing to practice a highly effective method of birth control for at least 4 weeks prior to randomization, and had to be willing to continue contraception until at least 4 weeks after the last dose of study treatment.
  3. Participants with chronic renal failure on dialysis（hemodialysis/ peritoneal dialysis） for ≥ 3 months prior to randomization，and that the frequency of dialysis was stable and no change in dialysis pattern was observed during the trial.
  4. On ESAs treatment for ≥8 weeks prior to screening stage with stable doses and the average doses ≤ 10000 IU/week. And two consecutive hemoglobin values ≥10.0 g/dL and ≤12.0 g/dL within 4 weeks prior to randomization.
  5. At least one transferrin saturation (TSAT) ≥ 20% and one serum ferritin (SF) level ≥ 100 ng/ml within 4 weeks prior to randomization. At least one serum folate level and vitamin B12 level ≥ lower limit of normal during the 4 weeks prior to randomization.
  6. Patient was informed of the investigational nature of the study and had given written, informed consent in accordance with institutional, local, and national guidelines.

Exclusion Criteria:

* Subjects who meet any of the following exclusion criteria are not to be enrolled in this study:

  1. Females who were pregnant or breast-feeding.
  2. Red blood cell (RBC) or whole blood transfusion within 12 weeks prior to randomization.
  3. Known intolerance to any ESA, parenteral iron supplementation, or PEGylated molecule.
  4. Known hematological disease (including but not limited to myelodysplastic syndrome, hematological malignancy, hemoglobinopathy, pure red cell aplasia, hemolytic syndromes, coagulation disorder, etc.) or cause of anemia other than renal disease（e.g. gastrointestinal bleeding or hookworm disease for stool occult blood positive，etc.）.
  5. Known autoimmune diseases（e.g. rheumatoid arthritis, systemic lupus erythematosus, anti-neutrophil cytoplasmic antibody related vasculitis, etc.）.
  6. Obvious infection occurred within 4 weeks prior to randomization，per investigator's clinical judgment.
  7. Chronic, uncontrolled, or symptomatic inflammatory disease，per investigator's clinical judgment.
  8. Uncontrolled or symptomatic secondary hyperparathyroidism，per investigator's clinical judgment.
  9. Poorly controlled hypertension within 4 weeks prior to randomization, per investigator's clinical judgment.
  10. Chronic congestive heart failure (New York Heart Association Class III~IV).
  11. Active hepatitis or any of the following check exceptions: ALT≥ 2 × upper limit of normal (ULN), AST≥ 2 × upper limit of normal (ULN), DBIL≥ 2 × upper limit of normal (ULN).
  12. A positive test for HIV antibody.
  13. Tumor malignancy（non-melanoma skin cancer and carcinoma in situ that have been resected are excluded）.
  14. Significant symptoms or diseases within 6 months prior to randomization，and the investigator judged that these diseases or symptoms may affect evaluation or follow-up.
  15. Expected survival less than 12 months.
  16. Planed to participate in a kidney transplant or have a kidney donor during the trial.
  17. Elective surgery during the study.
  18. Expected conception within 4 weeks after the end of the study treatment.
  19. The subject has participated in other clinical trial within the 12 weeks prior to randomization and throughout the trial period.
  20. Have any other condition or prior therapy that, in the investigator's opinion, would make the subject unsuitable for the study, or unable or unwilling to comply with the study procedures.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 372 (Actual)
Dates: Start 2019-05-15 (Actual); Primary Completion 2021-02-28 (Actual); Study Completion 2022-05-30 (Actual)

PRIMARY OUTCOMES:
The mean change from the baseline hemoglobin level to the mean level during the evaluation period | Week 17-24
  The primary efficacy end point is the mean change from the baseline hemoglobin level to the mean level during the evaluation period. The baseline hemoglobin value is defined as the mean of three hemoglobin values: the 4 weeks and 2 weeks recent hemoglobin values taken prior to the day of randomization and the value obtained on the day of randomization. The mean hemoglobin during the evaluation period was calculated as the mean of all available hemoglobin values during that period. Hemoglobin measurements will be performed at baseline and thereafter every 2 weeks (for the dose adjustment and the evaluation periods) or every 4 weeks (for the extensional treatment period).

SECONDARY OUTCOMES:
Proportion of Patients Whose Hemoglobin Within ±1.0 g/dL of Baseline during the Evaluation Period | Week 17-24
  The hemoglobin value within ±1.0 g/dL of baseline is defined as the difference between the hemoglobin value and the baseline value in the 4 tests in the Evaluation Period was at least 3 times between 1.0g /dL. The Evaluation Period is defined as study weeks 17 through 24.
Mean Dose of Participants With Hemoglobin Within ±1.0 g/dL of Baseline during the Evaluation Period | Week 17-24
  Mean dose was calculated at least 3 times from measurements taken during the Evaluation Period (Week 17 to Week 24).
Percentage of Participants With Hemoglobin Within the Target Range of 10.0 to 12.0 g/dL During the Evaluation Period | Week 17-24
  The hemoglobin value within the target range of 10.0 to 12.0 g/dL during the evaluation period is defined as HGB values were between 10.0 and 12.0 g/dL in at least 3 of the 4 tests in the efficacy evaluation period.
Average Hemoglobin, RBC, hematokrit and reticulocytes change from baseline | Week 0-52
  The baseline hemoglobin value is defined as the mean of three hemoglobin values: the 4 weeks and 2 weeks recent hemoglobin values taken prior to the day of randomization and the value obtained on the day of randomization.

OTHER OUTCOMES:
Safety Outcome Measures: adverse events | Week 0-52
  The incidence of patients who reported serious adverse events (SAE)
Safety Outcome Measures: composite safety endpoint(CSE) | Week 0-52
  The incidence of patients with risk cardiovascular events, The CSE consisted of five events: death, stroke, myocardial infarction, and serious adverse events of congestive heart failure and unstable angina. An independent Clinical Endpoint Committee (CEC) was used to provide blinded adjudication of potential CSE events.
Safety Outcome Measures: antibody | Week 17-24
  The incidence of patients with antibody to Pegol-Sihematide.

CONTACTS AND LOCATIONS:
Overall Officials: Jianghua Chen, MD, Principal Investigator — The First Affiliated Hospital, Zhejiang University
Locations (1):
- The First Affiliated Hospital, Zhejiang University, Hangzhou, Zhejiang, China

REFERENCES:
- [Derived] Zhang P, Jiang Y, Xu C, Zhou L, Zheng H, Xie D, Guo M, Huang X, Lu G, Jiang H, Qiu H, Liu B, Li S, Chen Q, Xia Y, Sun B, Yang X, Zhang S, Du S, Sun M, Chen M, Zhong A, Wang X, Zhao Z, Zhou H, Li G, Ren Y, Luo Q, Yang A, Luo P, Tang S, Xu C, Wang Q, Wang X, Yan T, He W, Qin S, Zhang W, Lv L, Wang C, Liu H, Li J, Wu Q, Pan C, Li C, He L, Chen J. Pegmolesatide for the treatment of anemia in patients undergoing dialysis: a randomized clinical trial. EClinicalMedicine. 2023 Oct 28;65:102273. doi: 10.1016/j.eclinm.2023.102273. eCollection 2023 Nov. PMID 37954906